CLINICAL TRIAL: NCT03688464
Title: Efficacy of Melatonin and Diphenhydramine Versus Placebo in Treatment of Nighttime Pruritus in Atopic Dermatitis
Brief Title: Treatment of Nighttime Pruritus in Atopic Dermatitis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study never started
Sponsor: University of Nebraska (Other)
Collaborators: Children's Hospital and Medical Center, Omaha, Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0197-18-FB
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Melatonin; Drugs, Generic; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Melatonin Treatment (Active Comparator): Subjects to receive melatonin 0.1 mg/kg (minimum dose of 1 mg, maximum dose of 5 mg) 30 minutes prior to bedtime (1 mg/ml oral compound suspension) for 4 weeks.
  Interventions: Drug: Melatonin
- Diphenhydramine Treatment (Active Comparator): Subject to receive diphenhydramine 2.5 mg/ml oral liquid, dosed at 1 mg/kg at bedtime for 4 weeks.
  Interventions: Drug: Diphenhydramine
- Placebo (Placebo Comparator): Subjects will receive cherry flavored placebo at bedtime for 4 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Melatonin — Drug to be administered for 4 weeks. Subjects will complete surveys prior to initiation and at the end of the study that will assess severity of eczema, quality of life, severity of itch, and sleep quality.
  Other Names: generic
  Arms: Melatonin Treatment
Drug: Diphenhydramine — Drug to be administered for 4 weeks. Subjects will complete surveys prior to initiation and at the end of the study that will assess severity of eczema, quality of life, severity of itch, and sleep quality.
  Other Names: Benadryl
  Arms: Diphenhydramine Treatment
Drug: Placebos — Drug to be administered for 4 weeks. Subjects will complete surveys prior to initiation and at the end of the study that will assess severity of eczema, quality of life, severity of itch, and sleep quality.
  Other Names: generic
  Arms: Placebo

SUMMARY:
This study will look at melatonin vs. first generation antihistamine vs. placebo in improving nighttime itching in children with atopic dermatitis.

DETAILED DESCRIPTION:
This will be a 6 week study to determine the efficacy of melatonin vs. first generation antihistamine vs. placebo in improving nighttime pruritus in children with atopic dermatitis.

Secondary aims will include:

1. Determine efficacy of melatonin vs. first generation antihistamine in management of sleep disturbance in children with atopic dermatitis
2. Compare differences between treatment groups in disease improvement
3. Compare differences between treatment groups in quality of life

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed eczema covering more than 5% of body surface area
* Ages 2-12 years old

Exclusion Criteria:

* Sleep disorder, including underlying insomnia
* Neuropsychiatric disorder
* Condition that requires use of antihistamines
* On systemic eczema therapy or monoclonal antibody for allergic diseases
* Unable to discontinue other antihistamine use
* Autoimmune disease as melatonin is contraindicated

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
POEM (Patient Oriented Eczema Measure) | 6 weeks
  This survey is a total of 7 questions that assesses the quality of life of patient's with eczema to determine their disease severity. The 7 questions are scored out of 4 points. A higher total score indicates a higher severity of disease.
EASI score | 6 weeks
  This tool is also used to assess severity of eczema. 4 different body regions are scored based on the percentage of eczema affecting the area. The calculations for each region are severity score x area score x known multiplier. A higher score indicates a higher severity of disease.

SECONDARY OUTCOMES:
5D Pruritus survey | 6 weeks
  This survey is a 5 question survey to assess severity of itch in patient's with eczema. The higher the score the worse the pruritus is and the more it affects the patient on a daily basis.
ESS-CHAD | 6 weeks
  This questionnaire is a series of questions that assesses sleepiness. Patient's can rank the situations based on a 3 point scale, 0 indicating would never doze and 3 indicating a high chance of dozing. A higher score indicates increased sleepiness.
Actigraphy | 6 weeks
  This device is worn on the wrist of a patient like a watch and records sleep-wake cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Kylie Liermann, DO, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No